CLINICAL TRIAL: NCT04368689
Title: The Feasibility and Examination of the Effects of Floatation-based Reduced Environmental Stimulation Therapy (REST) on a Community Sample With Posttraumatic Stress Disorder (PTSD)
Brief Title: The Feasibility and Examination of the Effects of Floatation-based REST on a Community Sample With PTSD
Acronym: FLOAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Terri deRoon Cassini, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00032660
Record Dates: First submitted 2020-04-01; First posted 2020-04-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: Floatation-based Reduced Environmental Stimulation Therapy; PTSD; FLOAT; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Floating (Experimental): Participants have 3 Floatation sessions that last up to 90 minutes. Each spaced about a week apart.
  Interventions: Other: Floatation-based reduced environmental stimulation therapy

INTERVENTIONS:
Other: Floatation-based reduced environmental stimulation therapy — Completion of 3 float session that can last for up to 90 minutes each session, each spaced approximately one week apart

SUMMARY:
This project is being done to explore the effects floating has on individuals who have a history of trauma with stress related symptoms.

DETAILED DESCRIPTION:
This pilot study looks to further the current floatation-based REST literature by exploring the therapy's effectiveness within a community-based sample of adults with PTSD. This type of sample allows the study the opportunity to recruit both veteran and civilian subjects, two populations that can suffer from this clinical diagnosis and stand to benefit from this therapy. This study will:

1. Evaluate the psychological effects of floating for a clinical, community sample with PTSD.
2. Evaluate the physiological effects of floating for a clinical, community sample with PTSD.
3. Evaluate the subjective effects of floating for a clinical, community sample with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Has posttraumatic stress disorder (PTSD) as confirmed by the PCL-5
* 18-60 years of age

Exclusion Criteria:

* History of neurological conditions (e.g., epilepsy, stroke, severe traumatic brain injury, Parkinson's disease, Alzheimer's disease or other forms of dementia)
* Any skin conditions or open wounds that could cause pain when exposed to saltwater
* Has floated previously
* Has Schizophrenia spectrum or other psychotic disorders
* Refuses to adhere to the Pre-Float Checklist
* Non-English speaking
* Inability to lay comfortably in a shallow pool of water
* Refuses participation in the floatation-REST sessions
* Refuses to sign the Float Liability Waiver prior to floating
* No Communicable disease (e.g.- HIV, Hepatitis A, B& C, tuberculosis, or measles)
* No psychoactive drugs or laxatives within the past week from scheduled float. Psychoactive drugs include, but are not limited to: methylenedioxymethamphetamine (MDMA), lysergic acid diethylamide (LSD), psilocybin, peyote, phencyclidine, ketamine).No recreational drug use (e.g.tetrahydrocannabinol,abuse of prescription medicine) day before or day of study visit. No antihistamine that causes drowsiness and no alcohol the day of the float sessions.
* Lack of control of bodily functions prior to scheduled float
* Fresh tattoos that would inhibit ability to float (consult with tattoo artist)
* Colored/dyed hair less than one week old from scheduled float
* Body tanning/spay/paint less than one week old from scheduled float
* Active suicidal ideation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Post Traumatic Stress Disorder (PTSD) symptom severity score as measured by Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline, week 2, week 3
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) A clinician-administered structured diagnostic interview that is considered the gold standard for assessing and diagnosing PTSD.
Change in Post Traumatic Stress Disorder (PTSD) symptom severity score as measured by PTSD Checklist for DSM-5 | Baseline, week 2, week 3
  PTSD Checklist for DSM-5 The PCL-5 consists of 20 items and it takes 5 to 10 minutes to administer. Participants are instructed to answer items based on their experience of symptoms since the trauma (hospitalization) or in the last month (1 month). Each item corresponds to a symptom in the DSM-5.
Change in depression symptom severity score as measured by the Center for Epidemiologic Studies Depression Scale - Revised | Baseline, week 2, week 3
  Center for Epidemiologic Studies Depression Scale - Revised Diagnostic tool for criteria for a major depressive episode
Change in depressive symptom severity score as measured by Patient Health Questionnaire (PHQ-9) | Baseline, week 2, week 3
  Patient Health Questionnaire (PHQ-9) The PHQ-9 is a 9-Item measure for assessing the severity of depressive symptoms over the past 2 weeks. Scores of 1-4 are considered indicative of minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.
Change in stress symptom score | Baseline, week 2, week 3
  Perceived Stress Scale The Perceived Stress Scale is a psychological instrument used for measuring an individual's perception of stress.
Change in Sheehan Disability Scale score | Baseline, week 2, week 3
  Sheehan Disability Scale How much mental health issues have affected their daily activities: work/school, social/leisure activities, and family life/home responsibilities. Total disability scores range between 0 to 30, with scores ≥ 5 signifying impairment.
Change in perceived happiness score | Baseline, week 2, week 3
  Fordyce Happiness Measure Measures emotional well being by perceived happiness
Change in anxiety symptom severity score | Baseline, week 2, week 3
  State-Trait Anxiety Inventory 20-item self-report questionnaire designed to assess an individual's level of anxiety.
Change in Positive and Negative Affect | Baseline, week 2, week 3
  Positive and Negative Affect Schedule - Expanded Form 20-items survey assessing general states of positive and negative affect using on a 5 point scale
Change in present moment sleepiness | Baseline, week 2, week 3
  Karolinska Sleepiness Scale Single item measure of present moment sleepiness
Change in pain score | Baseline, week 2, week 3
  Wong-Baker Pain scale Rates current level of pain from 0 to 10.
Change in Visual Analogue Scales score | Baseline, week 2, week 3
  Visual Analogue Scales- Relaxation, Muscle tension, Content/Peaceful, Refreshed, Energy & Overall Well-Being 7 measures rating on a 100-point scale and assessing overall well-being using a bipolar valence scale that goes from "Pretty Bad" to "Pretty Good"
Change in Side effect checklist score | Baseline, week 2, week 3
  Side effect checklist 43-item side effect checklist to assess the safety of Floatation- REST, and potential adverse experiences.
Change in Skin Conductance response post float | Baseline, Week 2, week 3
  Skin Conductance This will be measured using a program called "eSense". eSense (Mindfield Biosystems LLC), an ambulatory system for collecting skin conductance, or sweat gland activity. eSense samples skin conductance at 5 Hz, substantially lower than more traditional (and more expensive) laboratory systems. This will be done during the Trauma Narrative where subjects are asked to describe an event that they consider to be the most traumatic in their life including: who was there, what they were doing, where they were, how things looked, what they heard, etc.
Change in blood pressure post float | Baseline, Week 2, week 3
  -Blood Pressure This will be measured using a blood pressure cuff. This is performed before and after each float.
Change in number of mental health disorder diagnostic criteria met | Baseline, Week 3
  -Mini International Neuropsychiatric Interview - Depression (M.I.N.I. 7.0.2) The MINI is a short structured diagnostic interview designed to meet the need for a short but accurate psychiatric interview determining diagnostic criteria for 17 of the most common disorders in mental health. This version is for DSM-5 and ICD-10 diagnoses. The measure's psychometric properties of diagnostic validity and reliability have been determined to be strong
Anxiety sensitivity severity score pre float | Baseline
  -Anxiety Sensitivity Index (ASI-3) 18-item questionnaire using a 4-point scale and total ASI scores can range from 0 to 72. A meta-analysis [46] found that patient groups with anxiety and depression commonly have a total ASI score above 30, and other studies have used a cutoff score ≥ 30 to recruit individuals with very high levels of anxiety sensitivity.
Overall Anxiety Severity and Impairment score pre float | Baseline
  Overall Anxiety Severity and Impairment Scale A 5-item questionnaire that can be used across the different anxiety disorders as a continuous measure of anxiety severity and impairment over the past week. Each item is rated on a 5-point scale and the ratings are summed to obtain a total score ranging from 0 to 20.
Occurrence of adverse events post float | Week 3
  Debriefing Interview Occurrence of adverse events and qualitative information about floating. How was your float today? What did you think about while floating? Did anything surprise you? Did you learn anything about yourself?
  Follow-up Questions At the end of your float, how did you feel about the duration? Wanted to get out before/Perfect amount of time/Wish I could have stayed longer.
  Other techniques tried to help relax and feel less anxious and stressed? anti-anxiety medication/psychotherapy/massage/exercise/alcohol/breathing techniques/cigarettes/marijuana/progressive muscle relaxation/meditation/yoga/other Experience during and after today's float session compared to the other relaxation techniques tired? More relaxation with others/Equally as good as the others/More relaxation with floating than any others Interested in floating again in the future and thoughts on specialized pools being effective therapy for reducing symptom severity? Yes/No/Maybe

CONTACTS AND LOCATIONS:
Overall Officials: Terri deRoon-Cassini, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feinstein JS, Khalsa SS, Yeh HW, Wohlrab C, Simmons WK, Stein MB, Paulus MP. Examining the short-term anxiolytic and antidepressant effect of Floatation-REST. PLoS One. 2018 Feb 2;13(2):e0190292. doi: 10.1371/journal.pone.0190292. eCollection 2018. PMID 29394251
- [Background] Feinstein JS, Khalsa SS, Yeh H, Al Zoubi O, Arevian AC, Wohlrab C, Pantino MK, Cartmell LJ, Simmons WK, Stein MB, Paulus MP. The Elicitation of Relaxation and Interoceptive Awareness Using Floatation Therapy in Individuals With High Anxiety Sensitivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):555-562. doi: 10.1016/j.bpsc.2018.02.005. Epub 2018 Mar 9. PMID 29656950
- [Background] Fine TH, Turner JW Jr. The effect of brief restricted environmental stimulation therapy in the treatment of essential hypertension. Behav Res Ther. 1982;20(6):567-70. doi: 10.1016/0005-7967(82)90035-3. No abstract available. PMID 7159352
- [Background] Forgays, D. G., & Belinson, M. J. (1986). Is flotation isolation a relaxing environment?. Journal of Environmental Psychology, 6(1), 19-34.
- [Background] Jacobs GD, Heilbronner RL, Stanley JM. The effects of short term flotation REST on relaxation: a controlled study. Health Psychol. 1984;3(2):99-112. doi: 10.1037//0278-6133.3.2.99. PMID 6399246
- [Background] Kjellgren A, Sundequist U, Norlander T, Archer T. Effects of flotation-REST on muscle tension pain. Pain Res Manag. 2001 Winter;6(4):181-9. doi: 10.1155/2001/768501. PMID 11854763
- [Background] Koula, G. M., Kemp, J. C., Keane, K. M., & Belden, A. D. (1990). Replication of a clinical outcome study on a hospital-based stress management and behavioral medicine program utilizing flotation REST and biofeedback. In Restricted Environmental Stimulation (pp. 202-209). Springer, New York.
- [Background] Lilly, J.C. & Shurley, J.T. (1961).
- [Background] O'Leary, D. S., & Heilbronner, R. L. (1990). Flotation REST and information processing: A reaction time study. In Restricted Environmental Stimulation (pp. 113-124). Springer New York.
- [Background] Pudvah, M. B., & Rzewnicki, R. (1990). Six months in the tank: Long-term effects of flotation isolation on state anxiety, hostility, and depression. Restricted Environmental Stimulation: Theoretical and empirical developments in flotation REST, 169-173.
- [Background] Schulz P, Kaspar CH. Neuroendocrine and psychological effects of restricted environmental stimulation technique in a flotation tank. Biol Psychol. 1994 Mar;37(2):161-75. doi: 10.1016/0301-0511(94)90029-9. PMID 8003591
- [Background] Shurley, J. T. (1960). Profound experimental sensory isolation. American Journal of Psychiatry, 117(6), 539-545.
- [Background] Turner Jr, J., Gerard, W., Hyland, J., Nieland, P., & Fine, T. (1993). Effects of wet and dry flotation REST on blood pressure and plasma cortisol. In Clinical and Experimental Restricted Environmental Stimulation (pp. 239-247). Springer New York.